CLINICAL TRIAL: NCT03061500
Title: Proadrenomedullin as a Severity Score and Prognostic Marker in Intra-abdominal Sepsis
Brief Title: Prognostic Value of Proadrenomedullin in Intra-abdominal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Ana María Montero Fijoo, MD, Hospital Universitario La Paz
Other Study IDs: PI2289
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Intraabdominal Infections
Keywords: Proadrenomedullin; Sepsis; Intraabdominal Infections; prognosis
MeSH Terms: conditions — Intraabdominal Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational, prospective study whose main objective is to measure the value of Pro-adrenomedullin as a prognostic marker and predictor of mortality in patients with intra-abdominal sepsis after damage control surgery.

DETAILED DESCRIPTION:
Proadrenomedullin as a Severity Score and Prognostic Marker in Intra-abdominal Sepsis

Research Type:

Prospective, observational study.

Duration:

October 2016 - October 2017

Associated Medical Centers:

La Paz University Hospital (Madrid), La Princesa Hospital (Madrid), Hospital del Mar (Barcelona), Hospital Clínico de Valladolid and Hospital Clínico de Valencia.

Main Goal:

To measure the value of Pro-adrenomedullin as a prognostic marker and predictor of mortality in patients with intra-abdominal sepsis after damage control surgery.

Secondary Goals:

Make a comparison with other biomarkers (procalcitonin, lactic acid, CRP) and clinical severity scales used in standard critical practice (SAPSII, SOFA).

To establish a correlation between the levels of Pro-Adrenomedullin, the time of stay in critical care units, days of mechanical ventilation and mortality.

Variables:

A. Demographics

B. Date of admission to hospital and date of admission to critical care unit unit

C. Clinical data:

* Associated diseases
* SAPS II
* SOFA

D. Intra-abdominal infection episode data

* Systemic response: sepsis / septic shock
* Isolated microorganisms in blood cultures and intra-abdominal fluid
* Complications related to the infectious process (ARDS, need for mechanical ventilation, vasopressors, disseminated intravascular coagulation, acute renal failure, renal replacement techniques)

E. Follow-up

* Critical unit registration date
* Date of discharge from hospital
* Critical unit mortality, in-hospital mortality and 30 days mortality (assessed by telephone contact if the patient had been discharged).

F. Pro-adrenomedullin levels at admission, 24 and 72 hours. As well as procalcitonin (PCT), lactic acid and polymerase Chain Reaction (PCR) levels.

ELIGIBILITY:
Inclusion Criteria:

* All patients consecutively collected, adults over 18, who are admitted to critical care unit with the diagnosis of localized or generalized intraabdominal infection after damage control surgery.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with neutropenia induced by bone marrow transplant or by chemotherapy (<500 neutrophils / ml).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intraabdominal sepsis patients after damage control surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-10-15 (Estimated); Study Completion 2017-10-15 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days

SECONDARY OUTCOMES:
days of stay in critical units | 30 days
days of mechanical ventilation | 30 days
days of need vasopressors | 30 days
days of need for renal replacement techniques | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espana PP, Capelastegui A, Mar C, Bilbao A, Quintana JM, Diez R, Esteban C, Bereciartua E, Unanue U, Uranga A. Performance of pro-adrenomedullin for identifying adverse outcomes in community-acquired pneumonia. J Infect. 2015 May;70(5):457-66. doi: 10.1016/j.jinf.2014.12.003. Epub 2014 Dec 11. PMID 25499199
- [Background] Bello S, Lasierra AB, Minchole E, Fandos S, Ruiz MA, Vera E, de Pablo F, Ferrer M, Menendez R, Torres A. Prognostic power of proadrenomedullin in community-acquired pneumonia is independent of aetiology. Eur Respir J. 2012 May;39(5):1144-55. doi: 10.1183/09031936.00080411. Epub 2011 Nov 10. PMID 22075489
- [Background] Cavallazzi R, El-Kersh K, Abu-Atherah E, Singh S, Loke YK, Wiemken T, Ramirez J. Midregional proadrenomedullin for prognosis in community-acquired pneumonia: a systematic review. Respir Med. 2014 Nov;108(11):1569-80. doi: 10.1016/j.rmed.2014.09.018. PMID 25448309
- [Background] Suberviola B, Castellanos-Ortega A, Llorca J, Ortiz F, Iglesias D, Prieto B. Prognostic value of proadrenomedullin in severe sepsis and septic shock patients with community-acquired pneumonia. Swiss Med Wkly. 2012 Mar 19;142:w13542. doi: 10.4414/smw.2012.13542. eCollection 2012. PMID 22430899
- [Background] Christ-Crain M, Morgenthaler NG, Struck J, Harbarth S, Bergmann A, Muller B. Mid-regional pro-adrenomedullin as a prognostic marker in sepsis: an observational study. Crit Care. 2005;9(6):R816-24. doi: 10.1186/cc3885. Epub 2005 Nov 15. PMID 16356231